CLINICAL TRIAL: NCT06931418
Title: Randomized Controlled Trial for Post-operative Fracture Distal Radius Rehabilitation - The Early Motion Protocol Rehabilitation vs. Early Strengthening Study (EMPRESS Trial)
Brief Title: Early Strengthening Rehabilitation Training for Post-operative Fracture Distal Radius
Acronym: EMPRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Christian Xinshuo Fang, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 24-153
Record Dates: First submitted 2025-04-14; First posted 2025-04-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture; Rehabilitation; Patient outcomes; Physiotherapy; Occupational therapy; Orthopaedic fracture repair
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Double-blind randomised control trial with 50 patients in two interventional arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomly assigned to either one of the interventional arm and will not be informed of the randomisation result.
  Surgeons and assessors are blinded to the intervention allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Strengthening Protocol (ESP) (Experimental): Early use of strength and passive stretching will be encouraged after their initial assessment by rehabilitation therapists within 2 weeks of their discharge.
  Interventions: Other: Early Strengthening Protocol
- Early Motion Protocol (Control) (Active Comparator): Active mobilization is continued for the initial post-operative 6 weeks with allied health therapists, while passive mobilization and strengthening are started at the post-operative 8-10-week period.
  Interventions: Other: Early Motion Protocol

INTERVENTIONS:
Other: Early Strengthening Protocol — Patients in the ESP intervention arm will undergo active and passive exercises as well as strengthening exercises after their initial assessment by rehabilitation therapists within 2 weeks of their discharge. Early use of strength and passive stretching will be encouraged immediately after allocation.
  Arms: Early Strengthening Protocol (ESP)
Other: Early Motion Protocol — Patients are instructed for active flexion, extension, supination, pronation and finger flexion of the operated wrist along with motion of the shoulder and elbow after operation. Active mobilization is continued for the initial post-operative 6 weeks with allied health therapists. Passive mobilization and strengthening is started at the post-operative 8-10-week period.
  Arms: Early Motion Protocol (Control)

SUMMARY:
The primary objective of this study is to demonstrate safety and efficacy of an early strengthening and passive mobilization rehabilitation program for post-operative distal radius fracture fixation surgery compared to current conventional rehabilitation.

DETAILED DESCRIPTION:
Functional outcome after distal radius fracture fixation has often been variable with multiple factors affecting final results. Early mobilization rehabilitation protocols have been the gold standard after fracture fixation surgery. Rehabilitation protocols vary from center to center's own practices. However, these commonly encompass an early mobilization protocol or otherwise known as accelerated rehabilitation or enhanced recovery after surgery (ERAS) programs. Such programs comprise of a short duration of immobilization followed by a period of active mobilization before strengthening exercises are employed.

The investigators have performed early motion protocol (EMP) rehabilitation in the last decade in the investigation center for post-operative fracture distal radius fixation patients. The early motion protocol allows immediate active mobilization without a period of immobilization or splint protection. Despite early mobilization rehabilitation, there are a subset of patients who develop significant stiffness and pain with poor functional outcomes, especially in the early post-operative period. Moreover, some patients may also develop complex regional pain syndrome (CRPS) albeit early active mobilization. Thus, an early strengthening protocol (ESP) was developed to allow for immediate strengthening and passive mobilization exercises post-operatively with physiotherapist and occupational therapist guidance. Herein this study, the investigators hope to demonstrate the safety and efficacy of an ESP rehabilitation compared to EMP for post-operative distal radius fracture fixation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older
* Diagnosed with an isolated closed injury, displaced, distal radius fracture (AO/OTA Classification 23-A1-3, B1-2, C1-2) without articular comminution
* Requires operative fixation
* Able to give consent

Exclusion Criteria:

* History of previous hand or wrist surgery
* Neurological injury or pre-existing neurological conditions to the upper limb
* Underlying osteoarthritis of the wrist
* Unfit for surgical anesthesia
* Subacute fractures with delayed presentation (>2 weeks since initial injury)
* Unable to consent
* Refuse surgical intervention
* Unable to follow commands for rehabilitation
* Fixation construct or injuries requiring immobilization after surgery, such as unfixed distal ulna head or shaft fractures that require splintage or distal radio-ulnar joint instability planned for immobilization

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Region-specific patient reported functional outcome score | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Physical function and symptoms measured by Shortened Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH), an 11-item patient-reported measure with a total score ranging from 0 (no disability) to 100 (most severe disability).
Range of motion | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Subjects' wrist range of motion, including: pronation, supination, flexion, and extension will be measured by allied health therapists at each follow-up timepoint.
Grip strength | ESP group: At post-op weekly from 1 to 12 weeks, 6 months and 12 months ; EMP group: At post-op weekly from 6 to 12 weeks, 6 months and 12 months
  Grip strength will be measured using a dynamometer weekly for the ESP group and weekly from 6 weeks onwards for the EMP group.

SECONDARY OUTCOMES:
Health-related Quality of Life Measured by SF-12 Chinese (HK) Version | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  12-item Short Form Health Survey (SF-12), a patient-reported outcome measure of HRQOL comprised of a mental component (MCS) and physical component (PCS), each with a final score ranging from 0 (worst outcome) to 100 (best outcome).
Radiographic outcomes | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Subjects' X-rays will be assessed for fracture healing, implant migration, and fracture displacement.
Incidence of complications | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Incidence of wound breakdown, infection, CRPS, implant failure including screw breakage, and re-operation
Qualitative self-reported compliance | At post-op 2 weeks, 6 weeks , 12 weeks and 6 months and 12 months
  Subjects' self-reported score on their compliance to the rehabilitation exercises based on a Likert Scale of 1 (Did not follow) to 5 (Fully comply)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Prof. Fang, MBBS(HK), FRCS(Edinburgh), FHK, Principal Investigator — Dept of Orthopaedics and Traumatology, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset to be included as supplementary data in final publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year of study completion
Access Criteria: Additional information available upon reasonable request of principal investigator

REFERENCES:
- [Background] Tsutsui S, Kawasaki K, Yamakoshi K, Uchiyama E, Aoki M, Inagaki K. Impact of double-tiered subchondral support procedure with a polyaxial locking plate on the stability of distal radius fractures using fresh cadaveric forearms: Biomechanical and radiographic analyses. J Orthop Sci. 2016 Sep;21(5):603-8. doi: 10.1016/j.jos.2016.07.015. Epub 2016 Aug 12. PMID 27523260
- [Background] Baumbach SF, Synek A, Traxler H, Mutschler W, Pahr D, Chevalier Y. The influence of distal screw length on the primary stability of volar plate osteosynthesis--a biomechanical study. J Orthop Surg Res. 2015 Sep 8;10:139. doi: 10.1186/s13018-015-0283-8. PMID 26351239
- [Background] Ramavath A, Howard N, Lipscombe S. Biomechanical considerations for strategies to improve outcomes following volar plating of distal radius fractures. J Orthop. 2019 May 11;16(5):445-450. doi: 10.1016/j.jor.2019.04.006. eCollection 2019 Sep-Oct. PMID 31528050
- [Background] Handoll HH, Elliott J. Rehabilitation for distal radial fractures in adults. Cochrane Database Syst Rev. 2015 Sep 25;2015(9):CD003324. doi: 10.1002/14651858.CD003324.pub3. PMID 26403335
- [Background] Watson N, Haines T, Tran P, Keating JL. A Comparison of the Effect of One, Three, or Six Weeks of Immobilization on Function and Pain After Open Reduction and Internal Fixation of Distal Radial Fractures in Adults: A Randomized Controlled Trial. J Bone Joint Surg Am. 2018 Jul 5;100(13):1118-1125. doi: 10.2106/JBJS.17.00912. PMID 29975268
- [Background] Sorensen TJ, Ohrt-Nissen S, Ardenso KV, Laier GH, Mallet SK. Early Mobilization After Volar Locking Plate Osteosynthesis of Distal Radial Fractures in Older Patients-A Randomized Controlled Trial. J Hand Surg Am. 2020 Nov;45(11):1047-1054.e1. doi: 10.1016/j.jhsa.2020.05.009. Epub 2020 Jul 4. PMID 32636043
- [Background] Bhan K, Hasan K, Pawar AS, Patel R. Rehabilitation Following Surgically Treated Distal Radius Fractures: Do Immobilization and Physiotherapy Affect the Outcome? Cureus. 2021 Jul 7;13(7):e16230. doi: 10.7759/cureus.16230. eCollection 2021 Jul. PMID 34367829
- [Background] Andrade-Silva FB, Rocha JP, Carvalho A, Kojima KE, Silva JS. Influence of postoperative immobilization on pain control of patients with distal radius fracture treated with volar locked plating: A prospective, randomized clinical trial. Injury. 2019 Feb;50(2):386-391. doi: 10.1016/j.injury.2018.12.001. Epub 2018 Dec 4. PMID 30558805
- [Background] Blomstrand J, Kjellby Wendt G, Karlsson J, Wangdell J, Fagevik Olsen M. Pain, hand function, activity performance and apprehensiveness, in patients with surgically treated distal radius fractures. J Plast Surg Hand Surg. 2023 Feb-Dec;57(1-6):247-252. doi: 10.1080/2000656X.2022.2060992. Epub 2022 May 5. PMID 35510735
- [Background] Stinton SB, Graham PL, Moloney NA, Maclachlan LR, Edgar DW, Pappas E. Longitudinal recovery following distal radial fractures managed with volar plate fixation. Bone Joint J. 2017 Dec;99-B(12):1665-1676. doi: 10.1302/0301-620X.99B12.BJJ-2017-0348.R1. PMID 29212691
- [Background] Dillingham C, Horodyski M, Struk AM, Wright T. Rate of Improvement following Volar Plate Open Reduction and Internal Fixation of Distal Radius Fractures. Adv Orthop. 2011;2011:565642. doi: 10.4061/2011/565642. Epub 2011 Aug 11. PMID 21991417
- [Background] Sorensen AA, Howard D, Tan WH, Ketchersid J, Calfee RP. Minimal clinically important differences of 3 patient-rated outcomes instruments. J Hand Surg Am. 2013 Apr;38(4):641-9. doi: 10.1016/j.jhsa.2012.12.032. Epub 2013 Mar 6. PMID 23481405